CLINICAL TRIAL: NCT00003203
Title: An Intergroup Pilot Study of Concurrent Carboplatin, Vincristine and Radiotherapy Followed by Adjuvant Chemotherapy in Patients With Newly Diagnosed High-Risk Central Nervous System Embryonal Tumors
Brief Title: Carboplatin and Vincristine Plus Radiation Therapy Followed By Adjuvant Chemotherapy in Treating Young Patients With Newly Diagnosed CNS Embryonal Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A9971; COG-A9971 (Other: Children's Oncology Group); CCG-99701 (Other: Children's Cancer Group); CDR0000066055 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2003-05-19 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Brain Tumors; Central Nervous System Tumors; Neuroblastoma
Keywords: untreated childhood supratentorial primitive neuroectodermal tumor; untreated childhood medulloblastoma; localized unresectable neuroblastoma; regional neuroblastoma; stage 4S neuroblastoma
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Neoplasms; Neuroblastoma | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Carboplatin; Cisplatin; Cyclophosphamide; Vincristine; Chemotherapy, Adjuvant; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Newly diagnosed cerebral PNET with histologic verification (Experimental): Begin therapy within 31 days of surgery. Radiation therapy will be given in standard fractions along with filgrastim. The craniospinal axis will be treated first. Patients will receive carboplatin at 35 mg/m2/day IV over 15-20 minutes Monday through Friday, 1-4 hours prior to radiation for 6 weeks (total of 30 doses). Vincristine sulfate 1.5 mg/m2 IV will be given weekly x 6. Following radiation, patients will receive Maintenance chemotherapy. Patients enrolled prior to Amendment #5 will receive six cycles of cyclophosphamide and vincristine (Regimen A). Patients enrolled after Amendment #5 will receive six cycles of cyclophosphamide, vincristine sulfate and cisplatin (Regimen B).
  Interventions: Biological: filgrastim; Drug: carboplatin; Drug: cisplatin; Drug: cyclophosphamide; Drug: vincristine sulfate; Procedure: adjuvant therapy; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim — Given IV
  Other Names: G-CSF; Neupogen; NSC-614629
Drug: carboplatin — Given IV
  Other Names: Paraplatin; NSC-241240
Drug: cisplatin — Given IV
  Other Names: Platinol-AQ; NSC-119875
Drug: cyclophosphamide — Given IV
  Other Names: Cytoxan; NSC-26271
Drug: vincristine sulfate — Given IV
  Other Names: Oncovin; NSC-67574
Procedure: adjuvant therapy
Radiation: radiation therapy — 1.8 Gy/fx x 20fx=36Gy Craniospinal XRT*
  Other Names: radiotherapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin and vincristine, work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining carboplatin and vincristine with radiation therapy followed by adjuvant chemotherapy may kill more tumor cells.

PURPOSE: Randomized phase II trial to study the effectiveness of combination chemotherapy plus radiation therapy followed adjuvant chemotherapy in treating young patients who have newly diagnosed high-risk CNS embryonal tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasible dose and duration of carboplatin combined with craniospinal and local radiotherapy and adjuvant chemotherapy in children with newly diagnosed, high-risk CNS embryonal tumors (Phase I completed as of 11-25-03).
* Determine the feasibility of administering cyclophosphamide and vincristine with or without cisplatin after concurrent carboplatin, vincristine, and radiotherapy in these patients.
* Determine the overall and individual toxicity rates of this regimen in these patients.
* Determine the complete response rate in patients treated with this regimen.
* Obtain preliminary estimates of event-free survival of patients treated with this regimen.
* Determine the prognostic significance of enhancing tumor after completion of radiotherapy on event-free survival of these patients.

OUTLINE: This is a pilot, dose-escalation study of carboplatin. (Phase I completed as of 11-25-03.)

Within 31 days of definitive surgery, all patients receive vincristine IV weekly for 6 weeks and carboplatin IV over 15-20 minutes (after completion of vincristine infusion) 5 days a week for 6 weeks. Patients undergo radiotherapy (1-4 hours after carboplatin infusion) 5 days a week for 6 weeks.

Cohorts of 6-12 patients receive escalating doses of carboplatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 3 of 12 patients experience dose-limiting toxicity. (Phase I completed as of 11-25-03.)

At 6 weeks after completion of radiotherapy, patients are assigned to arm II for adjuvant/maintenance chemotherapy. (Arm I closed to accrual as of 11-25-03.)

* Arm I (closed to accrual as of 11-25-03): Patients receive cyclophosphamide IV over 1 hour on days 0 and 1, vincristine IV on days 0 and 7, and filgrastim (G-CSF) IV or subcutaneously (SC) beginning on day 2 and continuing for at least 10 days until blood counts recover.
* Arm II: Patients receive cyclophosphamide IV over 1 hour on days 1 and 2, vincristine IV on days 0 and 7, cisplatin IV over 6 hours on day 0, and G-CSF IV or SC beginning on day 3 and continuing for at least 10 days until blood counts recover.

In both arms, adjuvant/maintenance chemotherapy repeats every 4 weeks for 6 courses.

Patients are followed every 3 months for 8 months, every 4 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 162 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven high-risk CNS embryonal tumors, including:

  * Primitive neuroectodermal tumors
  * Atypical teratoid/rhabdoid tumor
  * Medulloblastoma
  * Desmoplastic medulloblastoma
  * Ependymoblastoma
  * Medullomyoblastoma
  * Spongioblastoma
  * Spongioblastoma polare
  * Primitive polar spongioblastoma
  * Neuroepitheliomatous neoplasms
  * Medulloepithelioma
  * Neuroblastoma
  * Pineoblastoma
* No bone marrow involvement or bone metastases
* No M4 disease
* M3 disease must have evidence of tumor on spinal MRI

PATIENT CHARACTERISTICS:

Age:

* 3 to 21 at diagnosis

Performance status:

* Not specified

Life expectancy:

* At least 8 weeks

Hematopoietic:

* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count at least 100,000/mm^3 (transfusion independent)
* Hemoglobin at least 10.0 g/dL (packed red blood cell transfusions allowed)

Hepatic:

* Bilirubin less than 1.5 mg/dL
* SGOT/SGPT less than 2.5 times normal

Renal:

* Creatinine less than 1.5 times upper limit of normal OR
* Creatinine clearance or radioisotope glomerular filtration rate at least 70 mL/min

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy

Surgery:

* Prior definitive surgery allowed

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 168 (Actual)
Dates: Start 1998-03; Primary Completion 2007-10 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Event Free Survival | Length of study
  Minimum time to disease progression or recurrence, time to death for any reason, or time to occurrence of a second malignant neoplasm (SMN).

SECONDARY OUTCOMES:
Survival | Length of study
  Time to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Regina Jakacki, MD, Study Chair — University of Pittsburgh
Locations (38):
- United States (35):
  - Long Beach Memorial Medical Center, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Children's Hospital of Denver, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Doernbecher Children's Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Grace Health Centre, Halifax, Nova Scotia

REFERENCES:
- [Result] Jakacki RI, Burger PC, Zhou T, Holmes EJ, Kocak M, Onar A, Goldwein J, Mehta M, Packer RJ, Tarbell N, Fitz C, Vezina G, Hilden J, Pollack IF. Outcome of children with metastatic medulloblastoma treated with carboplatin during craniospinal radiotherapy: a Children's Oncology Group Phase I/II study. J Clin Oncol. 2012 Jul 20;30(21):2648-53. doi: 10.1200/JCO.2011.40.2792. Epub 2012 Jun 4. PMID 22665539
- [Result] Jakacki R, Burger P, Zhou T, et al.: Outcome for metastatic (M+) medulloblastoma (MB) treated with carboplatin during craniospinal radiotherapy (CSRT) followed by cyclophosphamide (CPM) and vincristine (VCR): preliminary results of COG 99701. [Abstract] J Clin Oncol 25 (Suppl 18): A-2017, 2007.